CLINICAL TRIAL: NCT02464969
Title: A Randomized, Open-Label, Active Controlled, Safety and Descriptive Efficacy Study in Pediatric Subjects Requiring Anticoagulation for the Treatment of a Venous Thromboembolic Event
Brief Title: Apixaban for the Acute Treatment of Venous Thromboembolism in Children
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: B0661037; 2014-002606-20 (EudraCT Number); CV185-325 (Other: Alias Study Number)
Record Dates: First submitted 2015-05-26; First posted 2015-06-08 (Estimated); Results first posted 2024-10-29 (Actual); Last update posted 2024-10-29 (Actual); Status verified 2024-10

CONDITIONS: Venous Thromboembolism
Keywords: VTE, thromboembolism, thrombosis, embolism, apixaban, Eliquis
MeSH Terms: conditions — Venous Thromboembolism; Thromboembolism; Thrombosis; Embolism | interventions — apixaban; Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Apixaban (Experimental): Subjects between birth to <18 years will be dosed on a body weight tiered regimen. Subjects ≥35kg will receive 10mg twice daily(BID) for 7 days followed by 5mg BID thereafter;<35kg to 25kg will receive 8mg BID for 7 days followed by 4mg BID thereafter;<25 to 18kg will receive 6mg BID for 7 days and then 3mg BID thereafter;<18 to 12kg will receive 4mg BID for 7 days and then 2mg BID thereafter;<12 to 9kg will receive 3mg BID for 7 days and then 1.5mg BID thereafter;< 9kg to 6kg will receive 2 mg BID for 7 days and 1mg BID thereafter;<6kg to 5kg will receive 1mg BID for 7 days and 0.5mg BID thereafter;<5kg to 4kg will receive 0.6mg twice daily for 7 days and 0.3mg BID thereafter;PK cohort neonates ≥ 2.6kg will receive 0.1mg BID. Dose will be adjusted as determined by PK measurements (ie, to 0.2mg BID, 0.1mg daily or dose will stay the same).For the post PK cohort Neonates ˂4kg to 2.6kg, if confirmed by PK sub analysis,subjects will receive 0.2mg BID for 7 days and 0.1mg BID thereafter.
  Interventions: Drug: Apixaban; Drug: Standard of Care

INTERVENTIONS:
Drug: Apixaban — Tablet or Solution
Drug: Standard of Care — Unfractionated heparin, low molecular weight heparin, and/or a vitamin K antagonist. For subjects under 2 years of age, standard of care will be limited to unfractionated heparin or low molecular weight heparin.

SUMMARY:
To assess the safety and descriptive efficacy of apixaban in pediatric subjects requiring anticoagulation for the treatment of a VTE.

ELIGIBILITY:
Inclusion Criteria:

1. Birth to <18 years of age with a minimum weight of 2.6 kg at the time of randomization.
2. Presence of an index VTE which is confirmed by imaging.
3. Intention to manage the index VTE with anticoagulation treatment for at least 6 to 12 weeks.
4. Subjects able to tolerate oral feeding, nasogastric (NG), gastric (G) feeding and are currently tolerating enteric medications, as per investigator's judgement.

Exclusion Criteria:

1. Anticoagulant treatment for the index VTE for greater than 14 days prior to randomization. Neonates that are enrolled into the PK cohort must be on a minimum of 5 days and a maximum of 14 days SOC anticoagulation prior to randomization. Neonates that are enrolled into the post PK cohort may receive SOC anticoagulation for up to 14 days prior to randomization.
2. Thrombectomy, thrombolytic therapy, or insertion of a caval filter to treat the index VTE.
3. A mechanical heart valve.
4. Active bleeding or high risk of bleeding at the time of randomization.
5. Intracranial bleed, including intraventricular hemorrhage, within 3 months prior to randomization.
6. Abnormal baseline liver function at randomization.
7. Inadequate renal function at the time of randomization.
8. Platelet count <50×109 per L at randomization.
9. Uncontrolled severe hypertension at the time of randomization.
10. Use of prohibited concomitant medication at the time of randomization.
11. Female subjects who are either pregnant or breastfeeding a child.
12. Use of aggressive life-saving therapies such as ventricular assist devices (VAD) or extracorporeal membrane oxygenation (ECMO) at the time of enrollment.
13. Unable to take oral or enteric medication via the NG or G tube.
14. Known inherited or acquired antiphospholipid syndrome (APS).
15. Known inherited bleeding disorder or coagulopathy with increased bleeding risk (eg, hemophilia, von Willebrand disease, etc.)

Ages: 0 Days to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 229 (Actual)
Dates: Start 2015-11-22 (Actual); Primary Completion 2024-04-30 (Actual); Study Completion 2024-04-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (127):
- United States (83):
  - Pediatric Cardiology Clinic, Birmingham, Alabama
  - University of Alabama, Birmingham, Alabama
  - Phoenix Children's Hospital, Phoenix, Arizona
  - Loma Linda University Cancer Center, Loma Linda, California
  - Loma Linda University Children's Hospital, Loma Linda, California
  - Loma Linda University Medical Center, Loma Linda, California
  - Valley Children's Hospital, Madera, California
  - Children's Hospital and Research Center Oakland, Oakland, California
  - Bass Speicalty Pharmacy, Palo Alto, California
  - Inpatient Pharmacy, Palo Alto, California
  - Lucile Packard Children's Hosptial - Stanford University, Palo Alto, California
  - University of California Davis Comprehensive Cancer Center, Sacramento, California
  - Loma Linda University Health Care, San Bernardino, California
  - UCSF Benioff Children's Hospital, San Francisco, California
  - UCSF Mission Bay Pediatric Clinical Research Center, San Francisco, California
  - Children's Hospital Colorado - Investigational Drug Services, Aurora, Colorado
  - Children's Hospital Colorado, Aurora, Colorado
  - Connecticut Children's Medical Center Pharmacy, Hartford, Connecticut
  - Connecticut Children's Medical Center, Hartford, Connecticut
  - Nemours/ Alfred I. duPont Hospital for Children, Wilmington, Delaware
  - Childrens National Medical Center, Washington D.C., District of Columbia
  - UF Health Shands Hospital, Gainesville, Florida
  - JDCH Division of Pediatric Hematology and Oncology, Hollywood, Florida
  - Joe DiMaggio Children's Hospital, Hollywood, Florida
  - Memorial Regional Hospital, Hollywood, Florida
  - Nicklaus Children's Hospital, Miami, Florida
  - AdventHealth Orlando, Orlando, Florida
  - AdventHealth Orlando-Pharmacy Investigational Drug Services, Orlando, Florida
  - AdventHealth Pediatric Oncology Hematology at Orlando, Orlando, Florida
  - St. Joseph's Hospital, Tampa, Florida
  - Children's Hematology and Oncology a division of Kidz medical Service, West Palm Beach, Florida
  - St. Mary's Medical Center, West Palm Beach, Florida
  - Children's Healthcare of Atlanta-Egleston, Atlanta, Georgia
  - Children's Healthcare of Atlanta Center for Advanced Pediatrics - Pediatric Research Unit, Atlanta, Georgia
  - Children's Healthcare of Atlanta Center for Advanced Pediatrics-IDS Pharmacy, Atlanta, Georgia
  - Ann & Robert H Lurie Children's Hospital of Chicago, Chicago, Illinois
  - Bleeding and Clotting Disorders Institute, Peoria, Illinois
  - Unity Point Methodist Medical Center, Peoria, Illinois
  - OSF Saint Francis Medical Center, Peoria, Illinois
  - Indiana University, Indianapolis, Indiana
  - IU Health Pharmacy, Indianapolis, Indiana
  - Riley Hospital for Children at IU Health, Indianapolis, Indiana
  - University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - University of Kentucky Medical Center, Lexington, Kentucky
  - Boston Children's Hospital, Boston, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Children's Hospital of Michigan, Detroit, Michigan
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Children's Mercy Hospital, Kansas City, Missouri
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Columbia University Medical Center, New York, New York
  - New York-Presbyterian Morgan Stanley Children's Hospital, New York, New York
  - SUNY Upstate Medical University, Syracuse, New York
  - Levine Children's Specialty Center, Charlotte, North Carolina
  - Levine Children's Hospital, Pediatric Research, Charlotte, North Carolina
  - Levine Children's Hospital, Charlotte, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - Investigational Drug Service, Duke University Hospital, Durham, North Carolina
  - Sanford Children's Hospital, Fargo, North Dakota
  - Sanford Roger Maris Cancer Center, Fargo, North Dakota
  - Akron Children's Hospital, Akron, Ohio
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - University Hospitals Cleveland Medical Center, Cleveland, Ohio
  - Cleveland Clinic, Cleveland, Ohio
  - Nationwide Children's Hospital, Columbus, Ohio
  - OU Medical Center Investigational Drug Pharmacy, Oklahoma City, Oklahoma
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - The Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - St. Christopher's Hospital for Children, Philadelphia, Pennsylvania
  - UPMC Children's Hospital of Pittsburgh, Pittsburgh, Pennsylvania
  - Medical University of South Carolina: Investigational Drug Services, Charleston, South Carolina
  - Medical University of South Carolina: Shawn Jenkins Women's and Children's Hospital, Charleston, South Carolina
  - Medical University of South Carolina, Charleston, South Carolina
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Monroe Carell Jr. Children's Hospital at Vanderbilt, Nashville, Tennessee
  - Texas Children's Hospital- Main Hospital, Houston, Texas
  - Texas Children's Hospital- Wallace Tower, Houston, Texas
  - The Children's Hospital of San Antonio, San Antonio, Texas
  - University of Texas Health San Antonio, San Antonio, Texas
  - Primary Children's Hospital, Salt Lake City, Utah
  - Seattle Children's Hospital, Seattle, Washington
  - Children's Hospital of Wisconsin, Milwaukee, Wisconsin
  - Versiti Wisconsin, Milwaukee, Wisconsin
- Australia (3):
  - Kids Cancer Centre, Randwick, New South Wales
  - Prince of Wales Hospital, Sydney, New South Wales
  - The Royal Childrens Hospital, Parkville, VC
- Austria (3):
  - A.o.Landeskrankenhaus Innsbruck, Innsbruck, Tyrol
  - Medizinische Universitaet Innsbruck, Innsbruck
  - Medizinische Universitaet Wien, Vienna
- Canada (5):
  - Kaye Edmonton Clinic, Edmonton, Alberta
  - Stollery Children's Hospital, Edmonton, Alberta
  - Hamilton Health Science Corporation/McMaster Children's Hospital, Hamilton, Ontario
  - The Hospital For Sick Children, Toronto, Ontario
  - CHU Sainte-Justine, Montreal, Quebec
- France (5):
  - Hopital de la Timone Enfants, Marseille
  - CHRU de Montpellier - Hopital Arnaud de Villeneuve, Montpellier
  - Hopital Necker-Enfants malades, Paris
  - CHU de Bordeaux - Hopital Haut-Leveque, Pessac
  - Service d'Imagerie Medicale du Pr F. Laurent, Pessac
- Germany (3):
  - Charite - Universitaetsmedizin Berlin - Campus Virchow-Klinikum (CVK), Berlin
  - Universitätsklinikum Essen, Essen
  - Technische Universitat, Deutsches Herzzentrum Munchen, München
- Hadassah Medical Center (Ein Kerem), Jerusalem, Israel
- Mexico (2):
  - O.P.D Hospital Civil de Guadalajara, Hospital Civil Fray Antonio Alcalde, Guadalajara, Jalisco
  - Instituto Nacional De Cardiologia Ignacio Chavez, Mexico City
- Russia (3):
  - State Autonomous Healthcare Institution "Children's Republican Clinical Hospital of Ministry of, Kazan', Republic Tatarstan
  - State Autonomous Healthcare Institution of Sverdlovsk Region, Yekaterinburg, Sverdlovsk Oblast
  - FSBI "NRMC PHOI n.a.Dmitry Rogachev" of Minzdrav Russia, Moscow
- Spain (4):
  - Hospital Sant Joan de Deu, Esplugues de Llobregat, Barcelona
  - Hospital Universitario HM Monteprincipe, Boadilla del Monte, Madrid
  - Hospital Universitario Vall d´Hebron, Barcelona
  - Hospital Universitario La Paz, Madrid
- Turkey (Türkiye) (5):
  - Adana Acibadem Hospital, Seyhan, Adana
  - Baskent Universitesi Tip Fakultesi Cocuk Sagligi ve Hastaliklari ABD Cocuk Hematoloji Onkoloji BD, Bahçelievler, Ankara
  - Hacettepe University Faculty of Medicine, Ihsan Dogramaci Children's Hospital, Ankara
  - Ankara City Hospital Pediatric Hematology and Oncology Clinic, Ankara
  - Ege Universitesi Tip Fakultesi Cocuk Hastanesi Cocuk Hematoloji Bilim Dali, Izmir
- Ukraine (4):
  - Communal Enterprise "Dnipropetrovsk Specialized Clinical Medical Center of Mother and Child, Dnipro
  - Dnipropetrovsk Regional Children's Hospital, Dnipro
  - Municipal enterprise "Dnipropetrovsk Regional Children's Clinical Hospital", Dnipro
  - Communal Institution "Zaporizhzhia Regional Clinical Children's Hospital", Zaporizhzhia
- United Kingdom (6):
  - Royal Hospital for Children, Glasgow, Scotland
  - Newcastle Upon Tyne Hospitals NHS Foundation Trust, Newcastle upon Tyne, TYNE & WEAR
  - Cardiff & Vale NHS Health Board, Cardiff, Wales
  - Noah's Ark Children's Hospital for Wales, Cardiff, Wales
  - Birmingham Children's Hospital NHS Foundation Trust, Birmingham, WEST Midlands
  - Birmingham Women's and Children's NHS Foundation Trust, Birmingham, WEST Midlands

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=B0661037

RESULTS

PARTICIPANT FLOW:
Groups:
- Participants Receiving Apixaban: Participants between birth to <18 years were dosed on a body weight tiered regimen. Subjects ≥35kg received 10mg twice daily(BID) for 7 days followed by 5mg BID thereafter;<35kg to 25kg received 8mg BID for 7 days followed by 4mg BID thereafter;<25 to 18kg received 6mg BID for 7 days and then 3mg BID thereafter;<18 to 12kg received 4mg BID for 7 days and then 2mg BID thereafter;<12 to 9kg received 3mg BID for 7 days and then 1.5mg BID thereafter;< 9kg to 6kg received 2 mg BID for 7 days and 1mg BID thereafter;<6kg to 5kg received 1mg BID for 7 days and 0.5mg BID thereafter;<5kg to 4kg received 0.6mg twice daily for 7 days and 0.3mg BID thereafter; For sub group analysis, PK cohort neonates ≥ 2.6kg received 0.1mg BID. Dose was adjusted as determined by PK measurements (i.e., to 0.2mg BID, 0.1mg daily or dose stay the same).For the post PK cohort Neonates ˂4kg to 2.6kg, if confirmed by PK sub analysis ,participants received 0.2mg BID for 7 days and 0.1mg BID thereafter.
- Participants Treated With Standard of Care: Participants were treated with unfractionated heparin, low molecular weight heparin, and/or a vitamin K antagonist. For participants under 2 years of age, standard of care was limited to unfractionated heparin or low molecular weight heparin.
Period: Main Phase (Day 1 to Day 84)
Arm/Group | Participants Receiving Apixaban | Participants Treated With Standard of Care
Started | 155 | 74
Completed | 138 | 65
Not Completed | 17 | 9
Not completed — Adverse Event | 7 | 0
Not completed — Death | 1 | 1
Not completed — Lost to Follow-up | 3 | 0
Not completed — Withdrawal by Parent/Guardian | 0 | 4
Not completed — No Longer Meets Eligibility Criteria | 0 | 1
Not completed — Other Reasons | 4 | 2
Not completed — Entrance Criteria | 1 | 1
Not completed — Withdrawal by Subject | 1 | 0
Period: Extension Phase (Day 85 to Day 168)
Arm/Group | Participants Receiving Apixaban | Participants Treated With Standard of Care
Started | 53 (Participants who were earlier randomized to Apixiban group and clinically applicable continued in extension phase) | 0 (Participants randomized to SOC arm were not applicable to continue in extension phase.)
Completed | 50 | 0
Not Completed | 3 | 0
Not completed — Adverse Event | 1 | 0
Not completed — Withdrawal by Parent/Guardian | 1 | 0
Not completed — Other Reasons | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Participants Receiving Apixaban | Participants Treated With Standard of Care | Total
Number analyzed (Participants) | 155 | 74 | 229
Age, Continuous [Mean (Standard Deviation); unit: years] | 11.10 (6.51) | 11.68 (6.02) | 11.29 (6.35)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 85 | 43 | 128
  Male | 70 | 31 | 101
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 12 | 13 | 25
  Not Hispanic or Latino | 143 | 61 | 204
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 120 | 55 | 175
  Black | 22 | 9 | 31
  Asian | 5 | 4 | 9
  American Indian or Alaska Native | 1 | 0 | 1
  Other | 6 | 5 | 11
  Multiracial | 1 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Composite of Major and Clinically Relevant Non-Major (CRNM) Bleeding
Description: Bleeding definitions are based on the Perinatal and Paediatric Haemostasis Subcommittee of the International Society on Thrombosis and Haemostasis (ISTH) criteria. Major bleeding includes: (i) fatal bleeding; (ii) clinically overt bleeding with a decrease in Hgb of at least 20 g/L (2 g/dL) in 24 hours; (iii) retroperitoneal, pulmonary, intracranial, or central nervous system bleeding; and (iv) bleeding requiring surgical intervention in an operating suite (including interventional radiology). Clinically relevant non-major bleeding includes: (i) overt bleeding requiring a blood product not attributable to the participant's underlying condition; and (ii) bleeding requiring medical or surgical intervention to restore hemostasis, other than in an operating suite.
Time Frame: From first dose (Day 1) up to 114 days
Population: The safety data set (as-treated) consist of all randomized participants who received at least one dose of study drug. 95% CI was calculated using the Agresti-Coull method.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Participants Receiving Apixaban | Participants Treated With Standard of Care
Number analyzed (Participants) | 152 | 73
percentage of participants | 1.3 [0.1 to 5.0] | 1.4 [0.0 to 8.1]

2. Primary Outcome: Percentage of Participants With Symptomatic and Asymptomatic Recurrent Venous Thromboembolism (VTE) and VTE-Related Mortality
Description: Recurrent VTE, defined as either contiguous progression or non-contiguous new thrombus and including, but not limited to deep vein thrombosis (DVT), pulmonary embolism (PE) and paradoxical embolism. 95% CI was from the Agresti-Coull method.
Time Frame: From first dose (Day 1) up to 114 days
Population: The Full Analysis Set contains all randomized participants and also those assigned to apixaban post-protocol amendment 8.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Participants Receiving Apixaban | Participants Treated With Standard of Care
Number analyzed (Participants) | 155 | 74
percentage of participants | 2.6 [0.8 to 6.7] | 2.7 [0.2 to 9.9]

3. Secondary Outcome: Percentage of Participants Who Died
Description: Death due to any cause was assessed. 95% CI was calculated using the Agresti-Coull method.
Time Frame: From first dose (Day 1) up to 114 days
Population: The Full Analysis Set contains all randomized participants and also those assigned to apixaban post-PA8.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Participants Receiving Apixaban | Participants Treated With Standard of Care
Number analyzed (Participants) | 155 | 74
percentage of participants | 1.3 [0.1 to 4.9] | 1.4 [0.0 to 8.0]

4. Secondary Outcome: Percentage of Participants With Venous Thromboembolism (VTE)-Related Mortality
Description: Participants were assessed for death due to Venous Thromboembolism (VTE).
Time Frame: From first dose (Day 1) up to 114 days
Population: The Full Analysis Set contains all randomized participants and also those assigned to apixaban post-PA8.
Measure: Number; unit: percentage of participants
Arm/Group | Participants Receiving Apixaban | Participants Treated With Standard of Care
Number analyzed (Participants) | 155 | 74
percentage of participants | 0 | 0

5. Secondary Outcome: Number of Participants With Index Venous Thromboembolism (VTE) Status
Description: Index VTE status was defined as the last image obtained during the Main treatment phase for each participant's comparison to baseline imaging. Index VTE status was classified as Recurrence-contiguous; Recurrence-new; Unchanged; Regression; Resolution; Indeterminate/Nondiagnostic. Participants could have multiple concomitant index events. Regression was defined as (ie, unequivocal decrease [>50%] of the total volume/mass of the thrombus compared to the index event)
Time Frame: From first dose (Day 1) up to 91 days
Population: The Full Analysis Set contains all randomized participants and also those assigned to apixaban post-PA8. Excluding participants with a negative or Non-Diagnostic Index Event
Measure: Count of Participants; unit: Participants
Arm/Group | Participants Receiving Apixaban | Participants Treated With Standard of Care
Number analyzed (Participants) | 128 | 65
Participants
  Recurrence-contiguous | 2 | 0
  Recurrence-new | 0 | 0
  Unchanged | 8 | 6
  Regression | 25 | 11
  Resolution | 77 | 36
  Indeterminate/Nondiagnostic | 15 | 7
  Missing Follow-up Imaging, therefore cannot compare to baseline | 5 | 8
  Imaging not completed within the specified time period | 6 | 1

6. Secondary Outcome: Percentage of Participants With Stroke
Description: Participants were assessed for incidence of stroke.
Time Frame: From first dose (Day 1) up to 114 days
Population: The Full Analysis Set contains all randomized participants and also those assigned to apixaban post-PA8.
Measure: Number; unit: percentage of participants
Arm/Group | Participants Receiving Apixaban | Participants Treated With Standard of Care
Number analyzed (Participants) | 155 | 74
percentage of participants | 0 | 0

7. Secondary Outcome: Percentage of Participants With Symptomatic and Asymptomatic Recurrent Venous Thromboembolism (VTE)
Description: as for outcome 2
Time Frame: From first dose (Day 1) up to 114 days
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Participants Receiving Apixaban | Participants Treated With Standard of Care
Number analyzed (Participants) | 155 | 74
percentage of participants | 2.6 [0.8 to 6.7] | 2.7 [0.2 to 9.9]

8. Secondary Outcome: Number of Participants With New Symptomatic or Asymptomatic Deep Vein Thrombosis (DVT) and New Symptomatic or Asymptomatic Pulmonary Embolism (PE)
Description: Participants were assessed for incidence of Symptomatic or Asymptomatic Deep Vein Thrombosis (DVT) and New Symptomatic or Asymptomatic Pulmonary Embolism (PE).
Time Frame: From first dose (Day 1) up to 114 days
Population: The Full Analysis Set contains all randomized participants and also those assigned to apixaban post-PA8.
Measure: Count of Participants; unit: Participants
Arm/Group | Participants Receiving Apixaban | Participants Treated With Standard of Care
Number analyzed (Participants) | 155 | 74
Participants
  New Symptomatic or Asymptomatic DVT | 1 | 1
  New Symptomatic or Asymptomatic PE | 0 | 0

9. Secondary Outcome: Percentage of Participants With Other Symptomatic and Asymptomatic Venous Thromboembolism (VTE)
Description: Other VTE included events such as cerebral sinovenous thrombosis, renal vein thrombosis, portal vein thrombosis, catheter-related VTE, and splanchnic thrombosis. If VTE event type was blank, it was included in the Other VTE. 95% CI was from the Agresti-Coull method.
Time Frame: From first dose (Day 1) up to 114 days
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Participants Receiving Apixaban | Participants Treated With Standard of Care
Number analyzed (Participants) | 155 | 74
percentage of participants | 1.9 [0.4 to 5.8] | 1.4 [0.0 to 8.0]

10. Secondary Outcome: Number of Participants With Clinically Relevant Non-Major (CRNM) Bleeding, Major Bleeding and Minor Bleeding
Description: Bleeding definitions are based on the Perinatal and Paediatric Haemostasis Subcommittee of the International Society on Thrombosis and Haemostasis (ISTH) criteria. Major bleeding includes: (i) fatal bleeding; (ii) clinically overt bleeding with a decrease in Hgb of at least 20 g/L (2 g/dL) in 24 hours; (iii) retroperitoneal, pulmonary, intracranial, or central nervous system bleeding; and (iv) bleeding requiring surgical intervention in an operating suite (including interventional radiology). Clinically relevant non-major bleeding includes: (i) overt bleeding requiring a blood product not attributable to the participant's underlying condition; and (ii) bleeding requiring medical or surgical intervention to restore hemostasis, other than in an operating suite. Minor bleeding was defined as any overt or macroscopic evidence of bleeding that does not fulfill the above criteria for either major bleeding or clinically relevant, non-major bleeding.
Time Frame: From first dose (Day 1) up to 114 days
Population: The safety data set (as-treated) consist of all randomized participants who received at least one dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Participants Receiving Apixaban | Participants Treated With Standard of Care
Number analyzed (Participants) | 152 | 73
Participants
  Major Bleeding | 0 | 0
  Clinically Relevant Non-major Bleeding | 2 | 1
  Minor Bleeding | 54 | 21

11. Secondary Outcome: Blood Concentration of Apixaban (ng/mL)
Description: Blood samples were collected to assess the apixaban concentration at specified timepoints. Day 1 PK concentrations were only collected for participants in the Birth to ≤27 days arm. The lower limit of quantification (LLOQ) is 1.0 ng/mL for plasma samples, and 0.5 ng/mL for dried blood samples.
Time Frame: 3 hour (H), 12 H, 24 H at Day 3; pre and post dose at Day 14 and Day 42
Population: The PK analysis population is defined as all participants randomized to and treated with apixaban who have at least 1 concentration of apixaban. Participants with sample size of quantifiable values (≥ LLOQ) at the specified timepoints were analyzed.
Measure: Mean (Standard Deviation); unit: nanogram per millilitre (ng/mL)
Groups:
- Participants Between Age 12 to < 18 Years: Participants between age 12 to < 18 years were dosed on a body weight tiered regimen. Subjects ≥35kg received 10mg twice daily(BID) for 7 days followed by 5mg BID thereafter;<35kg to 25kg received 8mg BID for 7 days followed by 4mg BID thereafter;<25 to 18kg received 6mg BID for 7 days and then 3mg BID thereafter;<18 to 12kg received 4mg BID for 7 days and then 2mg BID thereafter;<12 to 9kg received 3mg BID for 7 days and then 1.5mg BID thereafter;< 9kg to 6kg received 2 mg BID for 7 days and 1mg BID thereafter;<6kg to 5kg received 1mg BID for 7 days and 0.5mg BID thereafter;<5kg to 4kg received 0.6mg twice daily for 7 days and 0.3mg BID thereafter.
- Participants Between Age 2 - < 12 Years: Participants between age 2 - < 12 years were dosed on a body weight tiered regimen. Subjects ≥35kg received 10mg twice daily(BID) for 7 days followed by 5mg BID thereafter;<35kg to 25kg received 8mg BID for 7 days followed by 4mg BID thereafter;<25 to 18kg received 6mg BID for 7 days and then 3mg BID thereafter;<18 to 12kg received 4mg BID for 7 days and then 2mg BID thereafter;<12 to 9kg received 3mg BID for 7 days and then 1.5mg BID thereafter;< 9kg to 6kg received 2 mg BID for 7 days and 1mg BID thereafter;<6kg to 5kg received 1mg BID for 7 days and 0.5mg BID thereafter;<5kg to 4kg received 0.6mg twice daily for 7 days and 0.3mg BID thereafter.
- Participants With Age 28 Days - < 2 Years: Participants with age 28 days - < 2 years were dosed on a body weight tiered regimen. Subjects ≥35kg received 10mg twice daily(BID) for 7 days followed by 5mg BID thereafter;<35kg to 25kg received 8mg BID for 7 days followed by 4mg BID thereafter;<25 to 18kg received 6mg BID for 7 days and then 3mg BID thereafter;<18 to 12kg received 4mg BID for 7 days and then 2mg BID thereafter;<12 to 9kg received 3mg BID for 7 days and then 1.5mg BID thereafter;< 9kg to 6kg received 2 mg BID for 7 days and 1mg BID thereafter;<6kg to 5kg received 1mg BID for 7 days and 0.5mg BID thereafter;<5kg to 4kg received 0.6mg twice daily for 7 days and 0.3mg BID thereafter.
- Participants in Age Group-Birth - ≤ 27 Days: Participants in age group-Birth - ≤ 27 days were dosed on a body weight tiered regimen. Subjects ≥35kg received 10mg twice daily(BID) for 7 days followed by 5mg BID thereafter;<35kg to 25kg received 8mg BID for 7 days followed by 4mg BID thereafter;<25 to 18kg received 6mg BID for 7 days and then 3mg BID thereafter;<18 to 12kg received 4mg BID for 7 days and then 2mg BID thereafter;<12 to 9kg received 3mg BID for 7 days and then 1.5mg BID thereafter;< 9kg to 6kg received 2 mg BID for 7 days and 1mg BID thereafter;<6kg to 5kg received 1mg BID for 7 days and 0.5mg BID thereafter;<5kg to 4kg received 0.6mg twice daily for 7 days and 0.3mg BID thereafter;PK cohort neonates ≥ 2.6kg received 0.1mg BID. Dose was adjusted as determined by PK measurements (ie, to 0.2mg BID, 0.1mg daily or dose stay the same).For the post PK cohort Neonates ˂4kg to 2.6kg, if confirmed by PK sub analysis ,participants received 0.2mg BID for 7 days and 0.1mg BID thereafter.
Arm/Group | Participants Between Age 12 to < 18 Years | Participants Between Age 2 - < 12 Years | Participants With Age 28 Days - < 2 Years | Participants in Age Group-Birth - ≤ 27 Days
Number analyzed (Participants) | 64 | 22 | 15 | 11
nanogram per millilitre (ng/mL)
  Hour 3 at Day 1: number analyzed (Participants) | 0 | 0 | 0 | 11
  Hour 3 at Day 1 |  |  |  | 30.7 (12.9)
  Hour 12 at Day 1: number analyzed (Participants) | 0 | 0 | 0 | 10
  Hour 12 at Day 1 |  |  |  | 13.9 (5.70)
  Hour 24 at Day 1: number analyzed (Participants) | 0 | 0 | 0 | 11
  Hour 24 at Day 1 |  |  |  | 23.3 (10.1)
  Pre-dose at Day 14: number analyzed (Participants) | 64 | 22 | 15 | 7
  Pre-dose at Day 14 | 61.1 (53.7) | 72.7 (42.5) | 56.4 (65.6) | 48.3 (23.0)
  Post-dose at Day 14: number analyzed (Participants) | 61 | 21 | 14 | 6
  Post-dose at Day 14 | 152 (80.2) | 189 (61.0) | 203 (118) | 119 (45.7)
  Pre-dose at Day 42: number analyzed (Participants) | 24 | 5 | 3 | 2
  Pre-dose at Day 42 | 54.5 (33.7) | 67.9 (33.8) | 123 (123) | 50.2 (34.1)
  Post-Dose at Day 42: number analyzed (Participants) | 27 | 7 | 4 | 3
  Post-Dose at Day 42 | 151 (79.1) | 212 (89.8) | 143 (88.0) | 109 (56.0)

12. Secondary Outcome: Concentration of Plasma Anti-Factor Xa (ng/mL)
Description: Blood samples were collected to assess the Anti-Factor Xa concentration at specified timepoints. Day 1 PK concentrations were only collected for participants in the Birth to ≤27 days arm. The lower limit of quantification (LLOQ) is 35.0 ng/mL.
Time Frame: Pre and post dose at Day 14 and Day 42
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: nanogram per millilitre (ng/mL)
Arm/Group | Participants Between Age 12 to < 18 Years | Participants Between Age 2 - < 12 Years | Participants With Age 28 Days - < 2 Years | Participants in Age Group-Birth - ≤ 27 Days
Number analyzed (Participants) | 60 | 20 | 13 | 3
nanogram per millilitre (ng/mL)
  Pre-dose at Day 14: number analyzed (Participants) | 51 | 18 | 10 | 3
  Pre-dose at Day 14 | 72.7 (60.4) | 82.7 (41.3) | 74.7 (69.7) | 48.0 (1.00)
  Post-dose at Day 14 | 147 (83.5) | 202 (75.8) | 190 (105) | 127 (4.04)
  Pre-dose at Day 42: number analyzed (Participants) | 20 | 4 | 2 | 0
  Pre-dose at Day 42 | 63.9 (27.4) | 75.3 (31.0) | 53.5 (13.4) |
  Post-Dose at Day 42: number analyzed (Participants) | 27 | 7 | 5 | 1
  Post-Dose at Day 42 | 153 (84.9) | 220 (98.4) | 156 (92.2) | 101 (NA) — Only 1 participant was analyzed hence SD not applicable

ADVERSE EVENTS:
Time Frame: Non-Serious adverse events were collected from first dose Day 1 up to end of treatment visit (Day 168) plus 35 days i.e., up to 203 days. Serious Adverse Events and all cause mortality was collected from Screening (Day -7) to end of treatment visit (Day 168) plus 35 days i.e., up to 210 days.
Description: Serious and non-serious adverse events were collected for safety population that includes all randomized participants who received at least one dose of study drug. All cause mortality was collected for all the randomized participants.
Arm/Group | Participants Receiving Apixaban | Participants Treated With Standard of Care
All-Cause Mortality (participants affected / at risk) | 2/155 | 1/74
Serious Adverse Events (participants affected / at risk) | 40/152 | 17/73
Other Adverse Events (participants affected / at risk) | 132/152 | 59/73
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Participants Receiving Apixaban (N=152) | Participants Treated With Standard of Care (N=73)
Cold type haemolytic anaemia (Blood and lymphatic system disorders) | 1 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 3 | 2
Myelosuppression (Blood and lymphatic system disorders) | 1 | 0
Neutropenia (Blood and lymphatic system disorders) | 1 | 0
Pancytopenia (Blood and lymphatic system disorders) | 1 | 0
Sickle cell anaemia with crisis (Blood and lymphatic system disorders) | 2 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 0
Cardiac arrest (Cardiac disorders) | 1 | 0
Cardio-respiratory arrest (Cardiac disorders) | 0 | 1
Cardiogenic shock (Cardiac disorders) | 1 | 0
Eye movement disorder (Eye disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0
Colitis (Gastrointestinal disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 1 | 0
Gastrointestinal pain (Gastrointestinal disorders) | 1 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 0
Haematemesis (Gastrointestinal disorders) | 1 | 0
Haematochezia (Gastrointestinal disorders) | 2 | 0
Ileus paralytic (Gastrointestinal disorders) | 1 | 0
Oesophagitis (Gastrointestinal disorders) | 1 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 1 | 0
Stomatitis (Gastrointestinal disorders) | 1 | 0
Chest pain (General disorders) | 0 | 1
Death (General disorders) | 1 | 0
Mucosal inflammation (General disorders) | 2 | 0
Multiple organ dysfunction syndrome (General disorders) | 1 | 0
Non-cardiac chest pain (General disorders) | 1 | 1
Peripheral swelling (General disorders) | 0 | 1
Pyrexia (General disorders) | 4 | 1
Drug-induced liver injury (Hepatobiliary disorders) | 1 | 0
Transplant rejection (Immune system disorders) | 1 | 0
Atypical pneumonia (Infections and infestations) | 1 | 0
Cellulitis (Infections and infestations) | 1 | 0
Device related bacteraemia (Infections and infestations) | 1 | 0
Escherichia pyelonephritis (Infections and infestations) | 0 | 1
Escherichia urinary tract infection (Infections and infestations) | 1 | 0
Gastroenteritis rotavirus (Infections and infestations) | 1 | 0
Infective pulmonary exacerbation of cystic fibrosis (Infections and infestations) | 1 | 0
Meningitis bacterial (Infections and infestations) | 1 | 0
Mycoplasma infection (Infections and infestations) | 1 | 0
Osteomyelitis (Infections and infestations) | 1 | 0
Pneumonia viral (Infections and infestations) | 1 | 0
Pseudomonal bacteraemia (Infections and infestations) | 1 | 0
Pyomyositis (Infections and infestations) | 0 | 1
Rhinovirus infection (Infections and infestations) | 1 | 0
Sepsis (Infections and infestations) | 1 | 0
Toxic shock syndrome (Infections and infestations) | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 0
Urinary tract infection bacterial (Infections and infestations) | 1 | 0
Varicella (Infections and infestations) | 0 | 1
Gun shot wound (Injury, poisoning and procedural complications) | 0 | 1
Incisional hernia (Injury, poisoning and procedural complications) | 0 | 1
Lower limb fracture (Injury, poisoning and procedural complications) | 1 | 0
Shunt thrombosis (Injury, poisoning and procedural complications) | 1 | 0
Suture rupture (Injury, poisoning and procedural complications) | 0 | 1
Alanine aminotransferase increased (Investigations) | 3 | 0
Blood urea increased (Investigations) | 0 | 1
Medical observation (Investigations) | 1 | 0
Weight increased (Investigations) | 1 | 0
Connective tissue disorder (Musculoskeletal and connective tissue disorders) | 1 | 0
Cytarabine syndrome (Musculoskeletal and connective tissue disorders) | 1 | 0
Embryonal rhabdomyosarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Cerebral venous sinus thrombosis (Nervous system disorders) | 2 | 0
Complex regional pain syndrome (Nervous system disorders) | 0 | 1
Headache (Nervous system disorders) | 0 | 1
Hypoxic-ischaemic encephalopathy (Nervous system disorders) | 0 | 1
Intracranial pressure increased (Nervous system disorders) | 1 | 0
Seizure (Nervous system disorders) | 0 | 1
Thoracic outlet syndrome (Nervous system disorders) | 1 | 0
Transient ischaemic attack (Nervous system disorders) | 0 | 1
Device malfunction (Product Issues) | 1 | 0
Depression (Psychiatric disorders) | 0 | 1
Munchausen's syndrome (Psychiatric disorders) | 0 | 1
Selective eating disorder (Psychiatric disorders) | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 1 | 0
Nephrotic syndrome (Renal and urinary disorders) | 1 | 0
Polyuria (Renal and urinary disorders) | 1 | 0
Heavy menstrual bleeding (Reproductive system and breast disorders) | 1 | 0
Acute chest syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hyperventilation (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumomediastinum (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Axillary vein thrombosis (Vascular disorders) | 1 | 0
Post thrombotic syndrome (Vascular disorders) | 1 | 0
Subclavian vein thrombosis (Vascular disorders) | 1 | 0
Superficial vein thrombosis (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Participants Receiving Apixaban (N=152) | Participants Treated With Standard of Care (N=73)
Anaemia (Blood and lymphatic system disorders) | 5 | 8
Leukopenia (Blood and lymphatic system disorders) | 3 | 4
Thrombocytopenia (Blood and lymphatic system disorders) | 5 | 4
Abdominal discomfort (Gastrointestinal disorders) | 0 | 4
Abdominal pain (Gastrointestinal disorders) | 11 | 5
Abdominal pain upper (Gastrointestinal disorders) | 8 | 4
Constipation (Gastrointestinal disorders) | 10 | 3
Diarrhoea (Gastrointestinal disorders) | 15 | 6
Nausea (Gastrointestinal disorders) | 12 | 5
Vomiting (Gastrointestinal disorders) | 22 | 4
Fatigue (General disorders) | 5 | 4
Injection site bruising (General disorders) | 1 | 12
Injection site haemorrhage (General disorders) | 0 | 4
Non-cardiac chest pain (General disorders) | 12 | 5
Pyrexia (General disorders) | 11 | 7
Upper respiratory tract infection (Infections and infestations) | 11 | 2
Contusion (Injury, poisoning and procedural complications) | 14 | 10
Hypokalaemia (Metabolism and nutrition disorders) | 3 | 4
Arthralgia (Musculoskeletal and connective tissue disorders) | 11 | 3
Back pain (Musculoskeletal and connective tissue disorders) | 8 | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 15 | 6
Headache (Nervous system disorders) | 27 | 10
Heavy menstrual bleeding (Reproductive system and breast disorders) | 16 | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 12 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 9 | 6
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 27 | 14
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 10 | 2
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 9 | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing, but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-04-28): https://cdn.clinicaltrials.gov/large-docs/69/NCT02464969/Prot_SAP_000.pdf